CLINICAL TRIAL: NCT07140354
Title: Regain of Arm and Hand Movements in Cervical Spinal Cord Injury Patients by Means of Spinal Transcutaneous Electrical Neuromodulation Assisted With an Arm Exoskeleton
Brief Title: Regain of Arm and Hand Movements in Cervical Spinal Stimulation
Acronym: tcSCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Guttmann (Other)
Responsible Party: Principal Investigator, Joan Vidal, Regain of arm and hand movements in cervical spinal cord injury patients by means of spinal electrical neuromodulation assisted with an arm exoskeleton., Institut Guttmann
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 235/C/2017
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injuries; cervical neuromodulation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tcSCS group (Experimental): The SCI individuals will receive transcutaneous Spinal Cord Stimulation (tcSCS) at the cervical level during upper extremity Ocupational therapy including ARMEO robotic therapy
  Interventions: Device: cervical transcutaneous spinal cord stimulation
- control group (Placebo Comparator): In the control group the SCI individuals will realize their routine ocupational therapy including ARMEO robotic therapywithout tSCS
  Interventions: Device: cervical transcutaneous spinal cord stimulation

INTERVENTIONS:
Device: cervical transcutaneous spinal cord stimulation — Cervical transcutaneous spinal cord stimulation (tSCS) delivers electrical currents over the cervical spinal cord to modulate neural circuits controlling the upper extremities. This approach has been shown to facilitate motor output, improve hand and arm function, and promote neuroplasticity in individuals with cervical spinal cord injury.

SUMMARY:
We will develop a "bottom to top" approach employing animal models and human testing to determine whether or not non-invasive neuro-modulation of the cervical spinal cord concomitant with upper limb rehabilitation driven by exo-skeletons can facilitate the regain of the arm and hand functional movements in spinal cord injured patients.

We hypothesize that that spinal electrical neuro-modulation together with sensory-motor rehabilitation will facilitate the transmission and processing of the motor commands along the residual brain-to-spinal connectome leading to the regain of arm and hand movements. The proposal follows a multi-disciplinary and translational approach; including basic scientists, engineers and clinicians, and is divided in 3 independent but related working packages (WP). WP1: Develop of a selfcontained hybrid robotic system to drive arm and hand movements rehabilitation in spinal cord injured patients. WP2: Implement the exo-skeleton to rehabilitate arm and hand movements concomitant to cervical electrical neuro-modulation in cervical spinal cord inured patients. WP3: In an animal model, using the optimal spinal stimulation parameters, identify the cellular and molecular changes in the brain-to-spinal connectome, which mediates recovery.

The results will support the development of the first feasible treatment to improve manual dexterity in cervical spinal cord inured patients, and will present a comprehensive and detailed analysis of the mechanisms underlying the recovery, providing an indispensable guideline for the application of stimulation-based therapy to SCI patients.

This proposal is a continuation of a recently awarded grant (2017-2020, funded by "Instituto Carlos III"), intended to obtain the optimal stimulation parameters to effectively neuromodulate the cervical spinal cord and facilitate arm function. The present proposal is the natural step forward, in which we want to explore in depth the mechanisms underpinning recovery, and further strength the rehabilitation intervention with arm exo

-skeleton, which will allow the performance of movements in severely injured patients.

DETAILED DESCRIPTION:
Patient selection criteria: The study will consist of two populations of patients: Population A will include a total of 10-15 patients with an incomplete cervical lesion (ASIA C and D), and a population B, with 8-15 patients with a complete motor cervical injury (ASIA A and B). Patients from both populations will have ages between 18 and 60 years, with a level of injury between C5 and T1 and with more than 12 months of evolution since the onset of the injury.

Experimental design:

Selected patients from both populations (A and B) will be included in one of the following groups: Group 1: Patients will receive conventional sensory-motor rehabilitation regimen of the upper limb concomitant; Group 2. Patients will receive conventional rehabilitation concomitant with transcutaneous electrical stimulation. Group 3: Patients will have exo-skeleton driven arm rehabilitation concomitant with transcutaneous electrical stimulation. Each session will last 40 minutes and will be done daily during the 6 weeks of evaluation.

Cervical transcutaneous stimulation protocol: Transcutaneous electrical stimulation will be applied by an external set of electrodes, which will be placed on the skin in the midline between the spinous processes of C6 and C8. Two rectangular plates (5.0 x 10.2 cm2) are placed on the skin of the shoulder blades and act as anodes. The electrical stimulation consist of monopolar pulse trains of 1 millisecond duration, released at a frequency of 10 kHz and at an intensity ranging from 80 to 180 mA. Each pulse train is presented at a frequency of 100Hz (ref 8). The stimulation intensity will be adjusted to 90% of the threshold to evoke contractions of the muscles. Rehabilitation of the upper limb. Conventional rehabilitation consists in voluntary, or assisted by a physical therapist, to manually articulate the upper extremities. Patients will perform motor and voluntary rehabilitation of the arms and hands to manipulate objects, performing exercises of grip, endurance and dexterity (ref 9) Robotic upper limb rehabilitation program.

By means of custom-made robotic exo-skeleton patients will move a joystick by a board, following a pattern presented on a television screen. The robot has a sensory feed back system, by which the regain of voluntary movements by the patients will decrease the force exerted by the exo-skeleton to move the arm. Patients will be included in the same number and length of sessions as the conventional rehabilitation regime. Neurological and functional evaluation. To evaluate the effectiveness of the intervention, prior to the initiation of rehabilitation, and once a month until the end of the study, a series of neurological, functional and daily life activities (ref 10) will be performed to evaluate the Effects of spinal stimulation on the motor control of the arms and hands. In addition, prior to the start and the end of each program, motor evoked potentials will be evaluated from the motor cortex and the monoand poly-synaptic reflexes evoked after peripheral nerve stimulation, in order to evaluate the acute and long-term changes in The cortico-medullary and own-medullary connectivity induced by the electrical stimulation.

Data analysis. Each patient will have previous and post-stimulation data. We will evaluate t-test between the different conditions, for each neurological and functional variable evaluated.

ELIGIBILITY:
Inclusion Criteria:

* male or female, more than 18 years old;
* a stable traumatic or no traumatic cervical SCI
* time since SCI: 3-12 months
* AIS A, B, C, and D with but at least ≥ 2 muscles affected in the upper extremities, with a total sum of muscle strength more than 2 points in two muscles (the wrist extension together with abductor pollicis brevis (APB) at least in one side).

Exclusion Criteria:

* unstable medical condition (cancer, acute infections, etc.)
* dependent on mechanical ventilation
* severe spasticity (≥3 score on the Modified Ashworth scale-MAS)
* contraindication for rehabilitation assisted with a robotic exoskeleton (Armeo®Power)
* peripheral nerve injury
* intolerance of tSCS, peacemakers, electronic implants, or episodes of epilepsy
* participating in another investigation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-09-08 (Actual)

PRIMARY OUTCOMES:
GRASSP | 2-3HRS
  The Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) is a standardized clinical tool designed to evaluate upper limb function in individuals with cervical spinal cord injury. It assesses strength, sensory function, and hand prehension ability to provide a comprehensive measure of hand and arm impairment.
MVC of upper extremity | 40-50MIN
  Maximum Voluntary Contraction (MVC) of the upper extremity refers to the greatest amount of force that a person can voluntarily generate with a specific muscle or muscle group of the arm or hand during an isometric contraction. It is commonly used as a standardized measure of muscle strength in research and rehabilitation, often recorded with devices such as dynamometers or force transducers.

SECONDARY OUTCOMES:
UEMS | 15-20min
  The Upper Extremity Motor Score (UEMS) is a component of the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) used to assess motor function in the upper limbs. It is calculated by testing five key muscle groups on each side (C5-T1), with scores ranging from 0 (total paralysis) to 5 (normal strength), for a maximum of 25 per side and 50 in total.
Spirometry for respiratory function | 20-30min
  Spirometry is a standardized pulmonary function test used to assess respiratory function by measuring airflow and lung volumes during forced breathing maneuvers. Key parameters include Forced Vital Capacity (FVC), Forced Expiratory Volume in 1 second (FEV₁), and the FEV₁/FVC ratio, which provide information on restrictive and obstructive ventilatory patterns.
MIP and MEP | 20-30min
  ChatGPT Plus
  Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP) are non-invasive measures of respiratory muscle strength.

OTHER OUTCOMES:
Quality of life measured by WhoQol-Bref | 20-30min
  Quality of life was measured by WhoQol-Bref based on a four-domain structure: physical health, psychological, social relationships, environment, and two questions about an individual's overall perception of their health.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Guttmann, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No